CLINICAL TRIAL: NCT02891798
Title: 4-drug Nerve Block Versus Plain Local Anesthetic for Knee and Hip Arthroplasty Analgesia in Veterans
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brian Williams (U.S. Federal Agency)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Brian Williams, VAPHS Surgical Specialties Service Line Medical Director, VA Pittsburgh Healthcare System
Organization: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO 1357; 13232002 (Other: USARMC)
Record Dates: First submitted 2016-08-12; First posted 2016-09-08 (Estimated); Results first posted 2021-12-20 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Pain
Keywords: analgesia,; buprenorphine; clonidine; dexamethasone; bupivacaine; nerve block
MeSH Terms: conditions — Pain; Agnosia | interventions — Bupivacaine; Clonidine; Buprenorphine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine + CBD (clonidine, buprenorphine, dexamethasone) (Experimental): Patients will receive a nerve block consisting of bupivacaine plus clonidine-buprenorphine-dexamethasone (Bupivacaine-CBD)
  Interventions: Drug: Bupivacaine + CBD (clonidine, buprenorphine, dexamethasone)
- Bupivacaine Only (control arm) (Active Comparator): Patients will receive a nerve block consisting of bupivacaine only.
  Interventions: Drug: Bupivacaine Only (control arm)

INTERVENTIONS:
Drug: Bupivacaine + CBD (clonidine, buprenorphine, dexamethasone) — Nerve blocks before surgery of L2-L4 and L4-S3 for Knee replacements Nerve blocks before surgery of L2-L4 for hip replacements
  Other Names: "Marcaine" + CBD (clonidine, buprenorphine, dexamethasone)
  Arms: Bupivacaine + CBD (clonidine, buprenorphine, dexamethasone)
Drug: Bupivacaine Only (control arm) — Nerve blocks before surgery of L2-L4 and L4-S3 for Knee replacements Nerve blocks before surgery of L2-L4 for hip replacements
  Other Names: Marcaine
  Arms: Bupivacaine Only (control arm)

SUMMARY:
After total joint replacement, early hospital discharge to home (with patients capable of continuing a home-based rehabilitation program) is a cost- effective management strategy. This project will use improved local anesthetic nerve block techniques to enhance technical capability and clinical practice by (i) reducing pain and other morbidities during recovery, (ii) improving weight-bearing achievement during in-hospital physical therapy to allow for earlier return home, and (iii) continued rehabilitation as an outpatient at home when feasible (versus in an extended care facility).

DETAILED DESCRIPTION:
Patients will have spinal anesthesia for their hip or knee replacement surgery. They will also receive the nerve blocks described above

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 85, and undergoing a total knee or hip replacement.
2. Fluent in English, decision competent, willing and able to provide written informed consent, and able to complete the study's schedule of assessments.
3. Able to walk >3m without an assisting device.
4. Have a BMI ≤ 40 kg/m2.

Exclusion Criteria:

1. Current participation in another orthopedic/Physical Therapy/rehab/anesthesiology interventional clinical trial.
2. Are at significant behavioral risks or have refractory major psychiatric disorders.
3. Revision surgery on the same extremity.
4. Have an American Surgical Association (ASA) Physical Status classification of 4 or higher.
5. Have been diagnosed with clinically significant neuropathy with its origins in either diabetes or other causes; have neuromuscular disease that would influence data collection.
6. Have a surgically-fused lumbar spine, or a spinal cord simulator, or other condition that would contraindicate or prohibit the conduct of spinal anesthesia.
7. At significant risk for postoperative substance abuse, or immediate-postoperative substance abuse withdrawal symptoms (alcohol, cocaine, enrolled in methadone or buprenorphine opioid withdrawal programs, etc.) Previous or current use of marijuana will not be an exclusion for study enrollment.
8. Are undergoing Total Knee Arthroplasty (TKA)/Total Hip Arthroplasty (THA) for a tumor.
9. Have contraindications (e.g., anaphylaxis) to any of the study drugs.
10. Have a systemic fungal infection.
11. Have a known hypersensitivity to bupivacaine hydrochloride or to any local anesthetic of the amide-type or to other components of bupivacaine hydrochloride solutions.
12. Have a known or suspected buprenorphine hypersensitivity (not including nausea and/or vomiting).
13. Have a gastro-intestinal (GI) obstruction.
14. Have paralytic ileus.
15. Pregnant women
16. Have had a kidney or liver transplant.

Veterans will not be excluded from participation based on smoking status, diagnosis of obstructive sleep apnea, or baseline monitored consumption of therapeutic opioids for documented medical indications; instead, these variables will be codified and quantified for subsequent covariate statistical analysis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2016-10; Primary Completion 2021-07-12 (Actual); Study Completion 2021-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Williams, MD, MBA, Principal Investigator — VA Pittsburgh Healthcare System
Locations (1):
- VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aloziem OU, Williams BA, Mikolic JM, Boudreaux-Kelly MY, Faruque S, Piva SR, Ibinson JW, Switzer GE. Assessing Common Content and Responsiveness of the QoR-15 and the SF-8 in the Context of Recovery from Regional Anesthesia for Joint Replacement. Mil Med. 2023 Nov 3;188(11-12):e3469-e3476. doi: 10.1093/milmed/usad191. PMID 37256753
- [Derived] Williams BA, Ibinson JW, Mikolic JM, Boudreaux-Kelly MY, Paiste HJ, Gilbert KL, Bonant SA, Ritter ME, Ezaru CS, Muluk VS, Piva SR. Day-One Pain Reductions After Hip and Knee Replacement When Buprenorphine-Clonidine-Dexamethasone Is Added to Bupivacaine Nerve/Plexus Blocks: A Randomized Clinical Trial. Pain Med. 2022 Jan 3;23(1):57-66. doi: 10.1093/pm/pnab325. PMID 34730810

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from November 2016 to October 2018 after HIPAA-compliant contact of the study recruiter by either the preoperative clinic or the orthopedic clinic clinical staff. Of the 571 screened, 473 were not eligible due to failing study inclusion/exclusion criteria (N=151), programmatic reasons (N=145), or not willing to participate (N=177), resulting in 98 patients enrolled in the study. Twenty of these were early terminations, leaving 78.
Pre-assignment Details: Study temporarily on-hold (6), Failed screening (3), Failed spinal (2), No study staff available (2), Surgery deferred (2), Current participation in another clinical trial (1), Intra-operative peri-prosthetic fracture (1), Patient chose another hospital (1), Surgery cancelled due to profuse vomiting after spinal anesthesia (1), and Uni-compartmental knee arthroplasty instead of total knee (1).
Groups:
- Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone): Patients will receive a nerve block consisting of bupivacaine plus buprenorphine-clonidine-dexamethasone (Bupivacaine-BCD)
  Bupivacaine + BCD (buprenorphine, clonidine, dexamethasone): Nerve blocks before surgery of L2-L4 and L4-S3 for Knee and hip replacements
- Bupivacaine Only (Control Arm): Patients will receive a nerve block consisting of bupivacaine only.
  Bupivacaine Only (control arm): Nerve blocks before surgery of L2-L4 and L4-S3 for Knee and hip replacements
Period: Overall Study
Arm/Group | Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) | Bupivacaine Only (Control Arm)
Started | 62 | 16
Completed | 62 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Veterans undergoing hip/knee replacement surgery completing the study course
Groups:
- Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone): Patients will receive a nerve blocks consisting of bupivacaine plus buprenorphine-clonidine-dexamethasone (Bupivacaine-BCD)
  Bupivacaine + BCD (buprenorphine, clonidine, dexamethasone): Nerve blocks before surgery of L2-L4 and L4-S3 for Knee and Hip replacements.
- Total: Total of all reporting groups
Arm/Group | Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) | Bupivacaine Only (Control Arm) | Total
Number analyzed (Participants) | 62 | 16 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (7.4) | 65.6 (7.6) | 66 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 56 | 13 | 69
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 53 | 15 | 68
  African American | 8 | 1 | 9
  Other | 1 | 0 | 1
  Hispanic | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62 | 16 | 78
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index
  kg/m^2 | 32.6 (4.6) | 31.9 (5.1) | 32 (5)
Diabetes [Number; unit: participants] | 23 | 6 | 29

OUTCOME MEASURES:

1. Primary Outcome: Short-Form McGill Pain Questionnaire (Version 2) Total Score Difference From Baseline
Description: SF-MPQ version 2 total score difference of Post-Operative Day 1 value minus the Baseline value. Differences can range from -10 to +10. Negative scores indicate a decrease in pain.
Time Frame: Baseline, Post-Operative day after surgery (7AM-9AM EST)
Population: All participants who completed the protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone): Patients will receive a nerve block consisting of bupivacaine plus buprenorphine-clonidine-dexamethasone (Bupivacaine-BCD)
  Bupivacaine + BCD (buprenorphine, clonidine, dexamethasone): Nerve blocks before surgery of L2-L4 and L4-S3 for Knee/Hip replacements
- Bupivacaine Only (Control Arm): Patients will receive a nerve block consisting of bupivacaine only.
  Bupivacaine Only (control arm): Nerve blocks before surgery of L2-L4 and L4-S3 for Knee/Hip replacements
Arm/Group | Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) | Bupivacaine Only (Control Arm)
Number analyzed (Participants) | 62 | 16
score on a scale | -1.85 (2.04) | -0.05 (2.38)
Statistical Analysis 1: Comparison: Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) vs Bupivacaine Only (Control Arm); Comparison of SF-MPQ2 Total Score Difference From Baseline between the 4-drug nerve block group and the bupivacaine only group; Test type: Superiority; p = 0.003, t-test, 2 sided

2. Primary Outcome: SF-MPQ2 Continuous Pain Subscore Difference From Baseline
Description: Continuous pain subscore difference of Post-Operative Day 1 value minus the Baseline value. Differences can range from -10 to +10. Negative scores indicate a decrease in pain.
Time Frame: Baseline, Post-Operative day after surgery (7AM-9AM EST)
Population: All participants who completed the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) | Bupivacaine Only (Control Arm)
Number analyzed (Participants) | 62 | 16
units on a scale | -2.29 (2.43) | 0.33 (2.76)
Statistical Analysis 1: Comparison: Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) vs Bupivacaine Only (Control Arm); Comparison of SF-MPQ2 Continuous Pain Subscore Difference From Baseline between the 4-drug nerve block group and the bupivacaine only group; Test type: Superiority; p = 0.001, t-test, 2 sided

3. Primary Outcome: SF-MPQ2 Intermittent Pain Subscore Difference From Baseline
Description: Intermittent pain subscore difference of Post-Operative Day 1 value minus the Baseline value. Differences can range from -10 to +10. Negative scores indicate a decrease in pain.
Time Frame: Baseline, Post-Operative day after surgery (7AM-9AM EST)
Population: All participants who completed the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) | Bupivacaine Only (Control Arm)
Number analyzed (Participants) | 62 | 16
units on a scale | -2.79 (2.66) | -1.14 (3.27)
Statistical Analysis 1: Comparison: Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) vs Bupivacaine Only (Control Arm); Comparison of SF-MPQ2 Intermittent Pain Subscore Difference From Baseline between the 4-drug nerve block group and the bupivacaine only group; Test type: Superiority; p = 0.038, t-test, 2 sided

4. Secondary Outcome: Quality of Recovery 15 Item Scale (QoR-15) Total Score
Description: Quality of Recovery 15 Item Scale, total score 0-150, 150 reflecting a perfect score and better recovery.
Time Frame: Day after surgery (7AM-9AM EST)
Population: All participants who completed the protocol. There was missing data for one participant in the Bupivacaine Only arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) | Bupivacaine Only (Control Arm)
Number analyzed (Participants) | 62 | 15
score on a scale | 106.08 (19.76) | 90.13 (24.15)
Statistical Analysis 1: Comparison: Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) vs Bupivacaine Only (Control Arm); Comparison of QoR-15 Total Score at post-operative day 1 between the 4-drug nerve block group and the bupivacaine only group; Test type: Superiority; p = 0.009, t-test, 2 sided

5. Secondary Outcome: Quality of Recovery 15 Item Scale (QoR-15) Total Score
Description: Quality of Recovery 15 Item Scale, total score 0-150, 150 reflecting a perfect score and better recovery.
Time Frame: 6 weeks post-operation
Population: All participants who completed the protocol. There was missing data for one participant in the Bupivacaine + BCD arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) | Bupivacaine Only (Control Arm)
Number analyzed (Participants) | 61 | 16
score on a scale | 128.89 (24.26) | 130.06 (21.75)
Statistical Analysis 1: Comparison: Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) vs Bupivacaine Only (Control Arm); Comparison of QoR-15 Total Score at 6 week post-procedure between the 4-drug nerve block group and the bupivacaine only group; Test type: Non-Inferiority — Testing the null hypothesis that Bupivacaine + BCD (buprenorphine, clonidine, dexamethasone) does not adversely affect recovery by producing a significantly lower score for the QoR-15 Total Score; p = 0.861, t-test, 2 sided

6. Secondary Outcome: Performed-based Physical Function is Assessed Using the Standing Balance Test.
Description: The Standing Balance Test score based on the ability of the participant to perform a series of standing exercises. Scores range from 0 to 4, with 4 indicating a longer time holding the stand (a better outcome).
  This test is germane to subjects with total joint replacement that are easily performed in the clinical settings. The test will capture the domains of muscle strength and activation, and balance.
Time Frame: 6 weeks post-operation
Population: All participants who completed the protocol. There was missing data for four participants in the Bupivacaine + BCD arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) | Bupivacaine Only (Control Arm)
Number analyzed (Participants) | 58 | 16
score on a scale | 3.86 (0.44) | 3.94 (0.25)
Statistical Analysis 1: Comparison: Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) vs Bupivacaine Only (Control Arm); Comparison of Standing Balance Test score at 6 week post-procedure between the 4-drug nerve block group and the bupivacaine only group; Test type: Non-Inferiority — Testing the null hypothesis that Bupivacaine + BCD (buprenorphine, clonidine, dexamethasone) does not adversely affect recovery by producing a significantly lower score for the Standing Balance test; p = 0.512, t-test, 2 sided

7. Secondary Outcome: Performed-based Physical Function is Assessed Using the Self-Selected Gait Speed Test.
Description: The Self-Selected Gait Speed Test is a timed test based on the ability of the participant to walk a 4 meter distance.
  This test is germane to subjects with total joint replacement that are easily performed in the clinical settings. The test captures the ability to walk.
Time Frame: 6 weeks post-operation
Population: All of the participants who completed the protocol. There was missing data for four participants in the Bupivacaine + BCD arm.
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) | Bupivacaine Only (Control Arm)
Number analyzed (Participants) | 58 | 16
meters per second | 0.88 (0.20) | 0.94 (0.21)
Statistical Analysis 1: Comparison: Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) vs Bupivacaine Only (Control Arm); Comparison of Self-Selected Gait Speed rate at 6 week post-procedure between the 4-drug nerve block group and the bupivacaine only group; Test type: Non-Inferiority — Testing the null hypothesis that Bupivacaine + BCD (buprenorphine, clonidine, dexamethasone) does not adversely affect recovery by producing a significantly slower rate for the Self-Selected Gait Speed test; p = 0.339, t-test, 2 sided

8. Secondary Outcome: Performed-based Physical Function is Assessed Using the Repeated Chair Stand Test.
Description: The Repeated Chair Stand Test is a timed test based on the ability of the participant to perform a series of standing exercises.
  This test is germane to subjects with total joint replacement that are easily performed in the clinical settings. The test will capture the domains of muscle strength and activation, and balance.
Time Frame: 6 weeks post-operation
Population: All participants who completed the protocol. There was missing data for five participants in the Bupivacaine + BCD arm.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) | Bupivacaine Only (Control Arm)
Number analyzed (Participants) | 57 | 16
seconds | 12.34 (4.31) | 11.93 (2.09)
Statistical Analysis 1: Comparison: Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) vs Bupivacaine Only (Control Arm); Comparison of Repeated Chair Stand time at 6 week post-procedure between the 4-drug nerve block group and the bupivacaine only group; Test type: Non-Inferiority — Testing the null hypothesis that Bupivacaine + BCD (buprenorphine, clonidine, dexamethasone) does not adversely affect recovery by producing a significantly slower time for the Repeated Chair Stand test; p = 0.711, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Throughout hospitalization, and at 2-week and 6-week postoperative visits.
Description: Adverse events reported here only include those that were unexpected in the normal course of surgery/anesthesia.
Groups:
- Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone): Patients will receive a nerve block consisting of bupivacaine plus buprenorphine-clonidine-dexamethasone (Bupivacaine-BCD)
  Bupivacaine + CBD (clonidine, buprenorphine, dexamethasone): Nerve blocks before surgery of L2-L4 and L4-S3 for Knee/Hip replacements
Arm/Group | Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) | Bupivacaine Only (Control Arm)
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/16
Other Adverse Events (participants affected / at risk) | 1/62 | 0/16
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine + BCD (Buprenorphine, Clonidine, Dexamethasone) (N=62) | Bupivacaine Only (Control Arm) (N=16)
Foot drop (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — One possibly block-related adverse event (foot drop after TKA), which resolved spontaneously over 4 months. The sciatic block for this patient was placed with ultrasound guidance; the intraoperative tourniquet time was 125 minutes (300 mmHg).

LIMITATIONS AND CAVEATS:
The sample size determined before the study began was N=100 patients to undergo primary THA and N=100 patients to undergo primary TKA, with these patients not undergoing physical therapy until day-one after surgery; these sample sizes were ultimately not achieved. By early 2018, same-day physical therapy (after surgery) became the new hospital guideline for patients undergoing primary THA and TKA, such that by mid-2018, the study was interrupted. Only the described 78 patients completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT02891798/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT02891798/ICF_001.pdf